CLINICAL TRIAL: NCT06823167
Title: A Phase 1 Study of IM-1021 in Participants With Advanced Malignancies
Brief Title: A Phase 1 Study of IM-1021 in Participants With Advanced Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Immunome, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IM-1021-101
Record Dates: First submitted 2025-02-04; First posted 2025-02-12 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Solid Malignancies; Hematologic Malignancies
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): IM-1021 administered intravenously on a 21-day cycle, at a starting dose of 2 mg/kg.
  Interventions: Biological: IM-1021

INTERVENTIONS:
Biological: IM-1021 — IM-1021 is an antibody-drug conjugate

SUMMARY:
IM-1021-101 is a Phase 1 study to determine the safety and effectiveness of IM-1021 in treating participants with advanced cancer.

DETAILED DESCRIPTION:
IM-1021-101 is a 2-part Phase 1 first-in-human (FIH), open-label, multicenter dose escalation and expansion study designed to determine the safety, tolerability, pharmacokinetics (PK), and preliminary anti-tumor activity of the ROR1 directed antibody-drug conjugate (ADC) IM-1021. IM-1021 will be administered to participants with advanced B-cell lymphomas and advanced solid tumors. Part A of the study is a dose escalation phase to evaluate safety and tolerability of IM-1021 and to determine recommended doses for further development. IM-1021 will be administered intravenously on an intermittent basis. The safety and tolerability of escalating doses of IM-1021 will be evaluated. Alternative dosing schedules may also be evaluated. Part B of the study is an expansion phase to further evaluate safety and tolerability of IM-1021 at candidate recommended doses in indication specific cohorts of participants. The safety and preliminary efficacy endpoints of this study will inform a preliminary risk-benefit assessment of IM-1021 in this patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent signed by the participant prior to conducting study-specific procedures
2. ≥18 years of age
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
4. Histological or cytological diagnosis of:

   Part A: advanced B-cell lymphomas or solid tumors, of the following subtypes:

   B-cell Lymphomas:
   * Mantle cell lymphoma (MCL)
   * Diffuse large B-cell lymphoma (DLBCL) (including Richter's transformation)
   * Follicular lymphoma
   * Small lymphocytic lymphoma (SLL)

   Solid Tumors:
   * Pancreatic cancer
   * Non-squamous non-small cell lung cancer (NSCLC)
   * Malignant mesothelioma
   * Epithelial ovarian cancer. Participants with fallopian tube and/or peritoneal malignancies are also eligible.
   * Triple-negative breast cancer.
   * Liposarcoma

   Other, unlisted histologies, if approved by the Sponsor Medical Monitor

   Part B Cohorts B1, B2, and B3:

   Histological or cytological diagnosis of the cohort-specific disease indication. Indications may include those listed in Inclusion Criterion 4.a
5. Participants must have adequate organ function.
6. Participants must have a negative pregnancy test, be willing to practice highly effective methods of birth control, use condoms, and refrain from oocyte/sperm donation, as applicable, as detailed in the protocol.
7. Participants must be refractory to or have relapsed after at least one prior standard therapeutic regimen. Participants must be relapsed or refractory to, have developed an intolerance to, or not be candidates for available therapies with established benefit. Participants with B-cell malignancies should have received at least two lines of therapy, including available therapies with established benefit. Participants with SLL should have received at least three prior lines of therapy.
8. Participants must have measurable disease as per the relevant response assessment framework: Lugano Classification for lymphoma (except SLL) , per iwCLL criteria for SLL , and per RECIST v.1.1 for solid tumors.

Exclusion Criteria:

1. Previously treated with an ADC with a topoisomerase-1 inhibitor payload, except: Participants with triple negative breast cancer may have received up to one prior ADC with a topoisomerase-1 inhibitor payload.
2. Previously received a ROR1-targeted therapy (eg, ADC, cell therapy, or monoclonal antibody).
3. History of an anaphylactic reaction to irinotecan or ≥ grade 3 GI toxicity to prior irinotecan.
4. Life expectancy < 12 weeks.
5. Prior solid organ transplant.
6. Participants with symptomatic ascites or pleural effusion. Participants who are clinically stable for at least 2 weeks following treatment for these conditions (including therapeutic thoraco- or paracentesis or catheter) are eligible.
7. Participant has a known active central nervous system (CNS) primary tumor or metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are clinically stable for at least 4 weeks prior to study entry, have no radiological evidence of new or enlarging brain metastases, and are off steroids or on a stable dose up to an equivalent of prednisone 10 mg/day for at least 15 days prior to first dose of study medication. Participants who have symptoms consistent with CNS metastasis must have a negative magnetic resonance imaging (MRI) or other clinically appropriate imaging study if the participant is not able to undergo contrast-enhanced MRI and approved by the Sponsor Medical Monitor during the screening period.
8. Participant has a known history of malignant primary brain tumor, or another primary solid or hematologic malignancy (other than that under study), unless the participant has undergone potentially curative therapy with no evidence of that disease for at least 2 years. Exception: The time requirement does not apply to participants who underwent successful definitive resection of certain cancers.
9. Participant has certain other significant medical conditions including cardiac, pulmonary, and infectious disease as detailed in the protocol.
10. Participant is pregnant, breastfeeding, or expecting to conceive within the projected duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of IM-1021 in participants with advanced lymphomas and advanced solid tumors as measured by incidence of treatment emergent adverse events (TEAEs) | From first dose to 37 days following last dose of study treatment
  Type, frequency, seriousness, and severity of adverse events (AEs) graded using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) criteria version 5.0, including serious adverse events (SAEs), AEs of interest (AEI), AEs leading to discontinuation, and deaths
Determine the recommended dose(s) and schedule(s) of IM-1021 for further development | From first dose to 37 days following last dose of study treatment
  Type, frequency, seriousness, and severity of adverse events (AEs) graded using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) criteria version 5.0, including serious adverse events (SAEs), AEs of interest (AEI), AEs leading to discontinuation, and deaths

SECONDARY OUTCOMES:
Area under the concentration-time curve (AUC) of IM-1021 in participants with advanced lymphomas and advanced solid tumors | Through 30-37 days following last dose of IM-1021 up to end of study
  Pharmacokinetic (PK) parameter
Concentration at end of infusion (Ceoi) of IM-1021 in participants with advanced lymphomas and advanced solid tumors | Through 30-37 days following last dose of IM-1021 up to end of study
  Pharmacokinetic (PK) parameter
Maximum observed concentration (Cmax) of IM-1021 in participants with advanced lymphomas and advanced solid tumors | Through 30-37 days following last dose of IM-1021 up to end of study
  Pharmacokinetic (PK) parameter
Time to maximum observed concentration (Tmax) of IM-1021 in participants with advanced lymphomas and advanced solid tumors | Through 30-37 days following last dose of IM-1021 up to end of study
  Pharmacokinetic (PK) parameter
Trough Concentration of IM-1021 in participants with advanced lymphomas and advanced solid tumors | Through 30-37 days following last dose of IM-1021 up to end of study
  Pharmacokinetic (PK) parameter
Apparent Terminal Half-Life (t1/2) of IM-1021 in participants with advanced lymphomas and advanced solid tumors | Through 30-37 days following last dose of IM-1021 up to end of study
  Pharmacokinetic (PK) parameter
Characterize the immunogenicity of IM-1021 | From first dose to about 30 days following last dose of study treatment
  Determined by the incidence of anti-drug antibodies (ADA) to IM-1021 from pre-infusion sample prior to each cycle.
To evaluate the preliminary anti-tumor activity of IM-1021 in participants with advanced lymphomas and advanced solid tumors | Week 6 until disease progression or participant discontinuation from study
  Objective response rate (ORR) as measured by Lugano Classification for participants with lymphoma (except SLL), per International Workshop on Chronic Lymphocytic Leukemia (iwCLL) criteria for participants small lymphocytic lymphoma (SLL), and per Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1 for participants with solid tumors
To evaluate the preliminary anti-tumor activity of IM-1021 in participants with advanced lymphomas and advanced solid tumors | Week 6 until disease progression or participant discontinuation from study
  Complete response rate (CRR) as measured by Lugano Classification for participants with lymphoma (except SLL), per International Workshop on Chronic Lymphocytic Leukemia (iwCLL) criteria for participants small lymphocytic lymphoma (SLL), and per Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1 for participants with solid tumors
To evaluate the preliminary anti-tumor activity of IM-1021 in participants with advanced lymphomas and advanced solid tumors | Week 6 until disease progression or participant discontinuation from study
  Disease control rate (DCR) as measured by Lugano Classification for participants with lymphoma (except SLL), per International Workshop on Chronic Lymphocytic Leukemia (iwCLL) criteria for participants small lymphocytic lymphoma (SLL), and per Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1 for participants with solid tumors

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - City Of Hope, Duarte, California
  - Yale University Medical Center, New Haven, Connecticut
  - University of Michigan, Ann Arbor, Michigan
  - START Midwest, Grand Rapids, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Gabrail Cancer Center, Canton, Ohio
  - Sarah Cannon Research Institute - Oncology Partners, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology, Irving, Texas

IPD SHARING:
Plan to Share IPD: Undecided